CLINICAL TRIAL: NCT00275028
Title: A Phase 2 Study of AZD2171 in Patients With Recurrent Ovarian, Primary Peritoneal Serous or Fallopian Tube Cancer
Brief Title: AZD2171 in Treating Patients With Recurrent Ovarian, Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00036; 05-170 (Other: Dana-Farber Cancer Institute); U01CA062490 (NIH)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2013-01

CONDITIONS: Fallopian Tube Cancer; Primary Peritoneal Serous Adenocarcinoma; Recurrent Ovarian Epithelial Cancer; Stage I Ovarian Epithelial Cancer; Stage II Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with recurrent ovarian, peritoneal, or fallopian tube cancer. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of AZD2171 in platinum sensitive and platinum insensitive disease, based on either RECIST criteria (for patients with measurable cancer radiographically) or clinical response benefit (modified Gynecologic Cancer Intergroup [GCIG] CA-125 response or stable disease for at least 16 weeks).

SECONDARY OBJECTIVES:

I. To assess progression-free survival. II. To assess modified GCIG CA-125 response rate. III. To assess duration of modified GCIG CA-125 response. IV. To assess the safety of the recommended phase 2 dose of AZD2171 in this asymptomatic patient population.

V. To explore the pharmacodynamic effects of AZD2171 by correlating clinical outcomes with an angiogenic profile derived from serial assessments of soluble VEGFR2, circulating endothelial cell levels, and VEGFR phosphorylation in circulating endothelial cells.

VI. To explore pharmacogenetic differences in kdr/flk-1, HIF1alpha, p53, and endothelial nitric oxide synthase (eNOS) in PBMCs from subjects who consent separately for pharmacogenetic studies.

VII. To determine whether oncogenic mutations predict response to AZD2171.

OUTLINE: This is a multicenter study. Patients are stratified according to disease sensitivity (platinum-sensitive disease vs platinum-insensitive disease).

Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* must have histologically or cytologically confirmed epithelial ovarian cancer, primary peritoneal serous cancer, or fallopian tube cancer
* must have either measurable cancer by RECIST criteria or an elevated CA125
* Subjects must be asymptomatic or minimally symptomatic
* Prior therapy:

  * Prior chemotherapy must have included a first-line platinum-based regimen only
  * Prior hormonal-based therapy for ovarian, primary peritoneal serous or fallopian tube cancer is acceptable
  * Up to two prior lines of chemotherapy in the recurrent setting are allowed
  * Toxic side effects related to prior chemotherapy or hormonal therapy must have resolved to less than or equal to grade 1 or to baseline (excluding alopecia), or for peripheral neuropathy to less than or equal to grade 2
  * Subjects may begin AZD2171 at least 3 weeks after their last dose of chemotherapy or hormonal therapy
* Life expectancy of greater than 6 months
* ECOG performance status 0-1 (Karnofsky >= 70%)
* must have lab values within normal institutional limits
* eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or PK of AZD2171 will be determined following review of their case by the Principal Investigator
* Subjects with treated limited stage basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the breast or cervix are eligible; subjects with stage I or II cancer treated with a curative intent are also eligible with no evidence of recurrent disease
* No evidence of preexisting uncontrolled hypertension; if patient has hypertension, it must be medically controlled
* AZD2171 has been shown to terminate fetal development in the rat, as expected for a process dependent on VEGF signaling; for this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry; must agree to use adequate contraception; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document- No therapeutic anticoagulation; the use of low dose warfarin (1 mg/day), intermittent doses of tPA (2 mg x 1), or heparin flushes to prophylax against central venous catheter-associated clots is permitted
* Measurable or non-measurable disease on CT scan or MRI
* Consider patients who have the following risk factors to be at increased risk; these patients should have increased monitoring:

  * Prior treatment with anthracyclines
  * Prior treatment with trastuzumab
  * A New York Heart Association classification of II controlled with treatment
  * Prior central thoracic radiation therapy (RT), including RT to the heart
  * History of myocardial infarction within 12 months

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or major surgery within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients may not be receiving any other investigational agents nor have participated in an investigational trial within the past 3 weeks; subjects may not have received prior treatment affecting the VEGF pathway; subjects may not have received prior treatment with antibodies that may interfere with CA-125 measurements; subjects may not have received intraperitoneal therapy within the 4 weeks prior to starting AZD2171 and/or the treating physician must confirm the patient has recurrent disease
* Patients may not be receiving any medication that may markedly affect renal function
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171
* Mean QTc > 500 msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome
* Uncontrolled intercurrent illness
* Pregnant women are excluded from this study because AZD2171 is a VEGF inhibitor with known abortifacient effects; breastfeeding should be discontinued if the mother is treated with AZD2171
* Major surgical procedure or medical interference with the peritoneum or pleura within 4 weeks of baseline CA-125 assessments
* Subjects with a history of an active malignancy during the last 3 years except non-melanomatous skin cancer , in situ breast or cervical cancer or stage I or II cancer treated with a curative intent and no active cancer recurrence
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2171
* No therapeutic anti-coagulation; prophylaxis against central venous catheter-associated clots is permitted
* A New York Heart Association classification of III or IV
* Conditions requiring concurrent use of drugs or biologics with proarrhythmic potentiate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-10; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Matulonis, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cediranib Maleate): Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cediranib maleate: Given orally
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate)
Started | 47
Completed | 0 (Participants are treated until one of the below milestones is reached. Completion is N/A.)
Not Completed | 47
Not completed — Withdrew consent before treatment began | 1
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 9
Not completed — Progressive Disease | 30
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: The number of patients analyzed reflects the intent-to-treat population.
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 56.5 [41 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White (non-Hispanic) | 45
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 46
Platinum Sensitivity [Number; unit: participants]
  Platinum Sensitive | 16
  Platinum Resistant | 30
Primary Cancer Diagnosis [Number; unit: participants]
  Ovarian cancer | 40
  Fallopian tube cancer | 1
  Peritoneal cancer | 5
Histologic Subtype [Number; unit: participants]
  Papillary serous | 38
  Endometrioid | 1
  Clear cell | 3
  Mixed type or other | 4
ECOG PS [Number; unit: participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS)
  0 - Normal activity.
  1. - Symptoms, but ambulatory.
  2. - In bed <50% of the time.
  3. - In bed >50% of the time.
  4. - 100% bed ridden.
  5. - Dead.
  participants
    0 | 34
    1 | 12
Tumor grade [Number; unit: participants]
  1 | 1
  2 | 0
  2-3 | 6
  3 | 39
Response Assessment [Number; unit: participants] — Refers to how the participants were followed for progression from baseline onward.
  participants
    RECIST | 36
    CA-125 | 10
Number of Prior Therapies for Recurrent Cancer [Number; unit: participants]
  0 | 19
  1 | 22
  2 | 5
Prior History of Hypertension [Number; unit: participants]
  Yes | 6
  No | 40

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Benefit (Modified Gynecologic Cancer InterGroup [GCIG] Cancer Antigen [CA]-125 Response or Stable Disease) Based on the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RESIST)
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 35
participants
  Stable Disease | 6
  Complete Response | 0
  Partial Response | 8
  Progressive Disease | 21

2. Secondary Outcome: Progression-free Survival
Time Frame: Up to 2 years
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 46
weeks | 18.43 (1.4278)

ADVERSE EVENTS:
Arm/Group | Treatment (Cediranib Maleate)
Serious Adverse Events (participants affected / at risk) | 17/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cediranib Maleate) (N=46)
CNS hemorrhage (Nervous system disorders) | 1
Rectal pain (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Small bowel obstruction (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Hypothermia (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hypertension (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cediranib Maleate) (N=46)
Diarrhea (Gastrointestinal disorders) | 42
Fatigue (General disorders) | 42
Hypertension (Cardiac disorders) | 36
Hypothyroidism (Endocrine disorders) | 26
Mucositis (Gastrointestinal disorders) | 24
Voice changes (Respiratory, thoracic and mediastinal disorders) | 21
Nausea (Gastrointestinal disorders) | 20
Headache (Nervous system disorders) | 22
Abdominal pain (Gastrointestinal disorders) | 21
Proteinuria (Renal and urinary disorders) | 10
Vomiting (Gastrointestinal disorders) | 16
Anorexia (Gastrointestinal disorders) | 9
Weight loss (Gastrointestinal disorders) | 8
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 6
Joint pain (Musculoskeletal and connective tissue disorders) | 6
Constipation (Gastrointestinal disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5
Muscle pain (Musculoskeletal and connective tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 12
ALT (Investigations) | 7
Alkaline phosphatase elevated (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 3
AST (Metabolism and nutrition disorders) | 6
Hot flashes (Vascular disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Urinary tract infection (Renal and urinary disorders) | 5
Fever (General disorders) | 3
Bloating (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 9
Chest pain (General disorders) | 4
Hemoglobin increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine increased (Investigations) | 3
Neuropathy (Nervous system disorders) | 15
Thrombocytopenia (Investigations) | 3
Oral pain (Gastrointestinal disorders) | 3
Hyperthyroidism (Endocrine disorders) | 4
Neutropenia (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less